CLINICAL TRIAL: NCT02688127
Title: Efficacy of Tranexamic Acid In Reducing Blood Loss Among Pregnant Women During Cesarean Section Because Of Placenta Previa
Brief Title: Efficacy of Tranexamic Acid In Reducing Blood Loss During Cesarean Section Because Of Placenta Previa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, shaimaa- sayed, Director , Clinical Research, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: r22wa2xt
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Postpartum Haemorrage Sever Bleeding After Delivery
Keywords: obstetric bleeding placenta previa
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tranexamic acid group (Experimental): tranexamic acid given as 1 gram intravenous dose dilute in 500 cc of ringer lactate 20 minute before cesarean section
  Interventions: Drug: Tranexamic Acid
- placebo group (Placebo Comparator): the control group will receive 500 cc of ringer lactate 20 minute before cesarean section
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — tranexamic acid or placebo are given before cesarean section in patient with placenta previa
  Other Names: cyclo kapron

SUMMARY:
This study evaluate role of tranexamic acid in reducing blood loss among pregnant women undergoing cesarean section because of placenta previa .Half of participants will receive tranexamia acid drug While the other half will receive placebo.

DETAILED DESCRIPTION:
Tranexamic Acid used in the field of obstetrics to decrease blood loss during and after cesarean section .

Tranexamic Acid is an antifibrinolytic agent which cause reversible and competitive blockade of the lysine binding sites in plasminogen molecules . It is a synthetic analog of amino acid lysine and its action is to reduce blood loss

ELIGIBILITY:
Inclusion Criteria:

* age 18 -38 Body mass index <30 , Diagnosis of placenta previa

Exclusion Criteria:

* patient with bleeding disorder , hepatic and renal disease. contraindication to tranexamic acid as allergy , hypersensitivity to tranexamic acid and known thromboembolic event during pregnancy .

other causes ofantepartum haemorrhage eg :accidental haemorrhage, rupture uterus.

type 1,2 of placenta previa anterior type 3,4 of placenta previa posterior causes of overdistended uterus like :multiple pregnancy, polyhydraminos

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Amount of Actual blood loss in each group | 6hour after operation
  observational

SECONDARY OUTCOMES:
Difference in haemoglobin before operation and 24 hours after operation | 24 hours
  observational

IPD SHARING:
Plan to Share IPD: Yes